CLINICAL TRIAL: NCT04422756
Title: Prospective Evaluation of Confirmatory Testing for Primary Aldosteronism
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Hypertension Canada (Other)
Responsible Party: Sponsor
Other Study IDs: REB16-2322
Record Dates: First submitted 2020-05-27; First posted 2020-06-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-07

CONDITIONS: Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Seated intravenous saline infusion test — The test will be conducted by infusing two litres of normal saline intravenously over 4 hours with the patient seated.Blood collection (for aldosterone, cortisol, renin, and electrolytes) will be performed at baseline and after completion of the infusion. Following infusion, plasma aldosterone levels <140 pmol/L will be considered as "negative," levels >280 pmol/L as "positive," and levels in between classified as indeterminate.
Diagnostic Test: Ultra low-dose ACTH stimulation test — The test will be performed by injecting 0.03 mcg of ACTH intravenously. Blood collection (for aldosterone, cortisol, and renin) will be performed at baseline and after 15 minutes. We expect a "positive" response to correspond with a plasma aldosterone >2200 pmol/L and ARR >220 pmol/L/mIU/L following stimulation.

SUMMARY:
This study is to evaluate the performance characteristics of the seated saline infusion test and the ultra low-dose ACTH stimulation test for the diagnosis of primary aldosteronism.

DETAILED DESCRIPTION:
This is a prospective study (with a target recruitment of 200 participants) designed to evaluate the performance characteristics of the seated saline infusion test and the ultra low-dose ACTH stimulation test for the diagnosis of primary aldosteronism, using disease-specific treatment response as a reference gold standard. Subjects consenting to study participation will undergo a standardized seated saline infusion test, followed by an ultra low-dose ACTH stimulation test. All participants also receive adrenal vein sampling. Individuals who have unilateral disease and desire surgery will receive adrenalectomy (as part of routine care) and the remaining subjects will receive medical treatment with a mineralocorticoid receptor antagonist. Response to targeted treatment will be considered the reference gold standard for the establishing the diagnosis of primary aldosteronism.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with hypertension
* Individuals with an elevated screening adrenal renin ration (ARR)
* Individuals with high probability features of primary aldosteronism (e.g., resistant hypertension, spontaneous or diuretic-induced hypokalemia, and/or an adrenal nodule) with clinical indications for adrenal vein sampling and surgery (if appropriate).

Exclusion Criteria:

* Individuals with chronic kidney disease (estimated glomerular filtration rate <40 mL/min/1.73m2),
* Individuals with a history of heart failure, chronic edema, uncontrolled severe hypertension (systolic blood pressure >180 and/or diastolic blood pressure >110 mmHg), untreated hypokalemia, cortisol-secreting adrenal adenoma, and/or pheochromocytoma
* Individual who previously received confirmatory testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertension individuals suspected of having primary aldosteronism.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of confirmatory testing (seated saline infusion test and the ultra low-dose ACTH stimulation test) | The total study timeline will occur over 66 months.
  Measures of diagnostic accuracy, as summarized by receiver operating characteristic curve analyses.

SECONDARY OUTCOMES:
The optimal cutoff value for confirmatory testing using clinically-important thresholds | The total study timeline will occur over 66 months.
  Plasma aldosterone
The optimal cutoff value for confirmatory testing using clinically-important thresholds | The total study timeline will occur over 66 months.
  Aldosterone-to-renin ratio

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Leung, Asst. Prof, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leung AA, Nerenberg K, Daskalopoulou SS, McBrien K, Zarnke KB, Dasgupta K, Cloutier L, Gelfer M, Lamarre-Cliche M, Milot A, Bolli P, Tremblay G, McLean D, Tobe SW, Ruzicka M, Burns KD, Vallee M, Prasad GV, Lebel M, Feldman RD, Selby P, Pipe A, Schiffrin EL, McFarlane PA, Oh P, Hegele RA, Khara M, Wilson TW, Penner SB, Burgess E, Herman RJ, Bacon SL, Rabkin SW, Gilbert RE, Campbell TS, Grover S, Honos G, Lindsay P, Hill MD, Coutts SB, Gubitz G, Campbell NR, Moe GW, Howlett JG, Boulanger JM, Prebtani A, Larochelle P, Leiter LA, Jones C, Ogilvie RI, Woo V, Kaczorowski J, Trudeau L, Petrella RJ, Hiremath S, Drouin D, Lavoie KL, Hamet P, Fodor G, Gregoire JC, Lewanczuk R, Dresser GK, Sharma M, Reid D, Lear SA, Moullec G, Gupta M, Magee LA, Logan AG, Harris KC, Dionne J, Fournier A, Benoit G, Feber J, Poirier L, Padwal RS, Rabi DM; CHEP Guidelines Task Force. Hypertension Canada's 2016 Canadian Hypertension Education Program Guidelines for Blood Pressure Measurement, Diagnosis, Assessment of Risk, Prevention, and Treatment of Hypertension. Can J Cardiol. 2016 May;32(5):569-88. doi: 10.1016/j.cjca.2016.02.066. Epub 2016 Mar 10. PMID 27118291
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Background] Mulatero P, Milan A, Fallo F, Regolisti G, Pizzolo F, Fardella C, Mosso L, Marafetti L, Veglio F, Maccario M. Comparison of confirmatory tests for the diagnosis of primary aldosteronism. J Clin Endocrinol Metab. 2006 Jul;91(7):2618-23. doi: 10.1210/jc.2006-0078. Epub 2006 May 2. PMID 16670162
- [Derived] Leung AA, Padwal RS, Hundemer GL, Venos E, Campbell DJT, Holmes DT, Orton DJ, So CB, Przybojewski SJ, Caughlin CE, Pasieka JL, Rabi DM, Kline GA. Seated Saline Suppression Test for Lateralizing Primary Aldosteronism. Hypertension. 2026 Jan 26. doi: 10.1161/HYPERTENSIONAHA.125.26008. Online ahead of print. PMID 41582811
- [Derived] Leung AA, Padwal RS, Hundemer GL, Venos E, Campbell DJT, Holmes DT, Orton DJ, So CB, Przybojewski SJ, Caughlin CE, Pasieka JL, Rabi DM, Kline GA. Confirmatory Testing for Primary Aldosteronism : A Study of Diagnostic Test Accuracy. Ann Intern Med. 2025 Jul;178(7):948-956. doi: 10.7326/ANNALS-24-03153. Epub 2025 May 6. PMID 40324193